CLINICAL TRIAL: NCT01039220
Title: Incidence of H1N1v Influenza-like Illness and Risk Factors for Serious Influenza Forms in HIV Infected Patients
Acronym: ANRS 2H
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Responsible Party: Name/Official Title: Lucie Marchand/Project manager, French National Agency for Research on AIDS and Viral Hepatitis
Organization: ANRS, Emerging Infectious Diseases (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2009-AO1115-52
Record Dates: First submitted 2009-12-22; First posted 2009-12-24 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2011-02

CONDITIONS: HIV Infections; Influenza
MeSH Terms: conditions — HIV Infections; Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: naso-pharyngeal swab — Selected patients will be asked to contact the clinical staff on site as soon as any influenza like symptoms appear. In the case of influenza like illness patients are requested to attend to the clinic within 24 hours for physical examination and naso-pharyngeal swab for diagnosis of A(H1N1)v infection.

SUMMARY:
To estimate the incidence of H1N1v influenza-like illness and to study the risk factors for serious influenza forms during pandemic period in French HIV infected patients.

* Definitions:

  * Influenza like illness is defined as fever> 37°8C and cough or pharyngalgia. (Centers for Disease Control definition).
  * Serious forms of influenza-like illness is defined by hospitalization within 14 days onset of symptoms or death attributed to influenza like illness.
* Design:

  * Survey sampling for estimating H1N1v influenza-like illness incidence.
  * Out of approximately 50 000 patients under follow-up in one of the 40 ANRS centres, a sub-group will be selected by random sampling. Sampling will be stratified by centre and sampling fraction per site will vary in order to select 60 to 80 patients for this study per site. A total of 2500 to 3000 patients will be selected to allow for estimating the incidence of H1N1v influenza-like illness with an adequate precision.

Selected patients will be asked to contact the clinical staff on site as soon as any influenza like symptoms appear. In the case of influenza like illness patients are requested to attend to the clinic within 24 hours for physical examination and naso-pharyngeal swab for diagnosis of A(H1N1)v infection.

Nested case-control study for the determination of risk factors for serious forms:

* Cases: Serious forms (see definition above) identified by any clinical site or hospitalisation unit.
* Controls: Patients of the randomly selected sample (see survey sampling above), presenting with influenza-like illness without any criterion for severity.

Exhaustivity check:

The exhaustivity of symptomatic forms will be assessed a posteriori by merging information from all available data sources.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Able to give written consent
* Covered by French Social Security
* HIV-infected (infection attested by the patient's chart)
* pregnant women

  * Control and sample to estimate incidence
* Patients followed for their HIV-infection in an ANRS center

  * Serious form
* Hospitalization whatever is the service in 14 days consecutive to a H1N1v influenza syndrome such as defined, or death consecutive to a H1N1v influenza syndrome such as defined.

Exclusion Criteria:

* patients for whom a H1N1v influenza syndrome can be informed at the beginning of the study.
* Under protection(saving) of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1266 (Actual)
Dates: Start 2009-12; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Serious forms (see definition above) identified by any clinical site or hospitalisation unit-Controls: Patients of the randomly selected sample (see survey sampling).

SECONDARY OUTCOMES:
Exhaustivity check: The exhaustivity of symptomatic forms will be assessed a posteriori by merging information from all available data sources.

CONTACTS AND LOCATIONS:
Overall Officials: Genevieve CHENE, Principal Investigator — INSERM U897 BORDEAUX
Locations (1):
- 34 ANRS center, Paris + Region of Country, France

REFERENCES:
- See also: (legal sponsor's website) — http://www.anrs.fr